CLINICAL TRIAL: NCT04157296
Title: Neurally Targeted Cognitive Training to Augment Cognitive Behavioral Therapy (CBT) Outcomes in Pediatric Anxiety
Brief Title: Neurally Targeted Cognitive Training to Augment CBT Outcomes in Pediatric Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Yanni Liu, Research Assistant Professor, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00169730; 5UL1TR002240-03 (NIH)
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Results first posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Anxiety Disorders
Keywords: anxious; Cognitive behavioral therapy; Computerized cognitive training
MeSH Terms: conditions — Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: A clinician, blind to whether patients are completing CCT or not, will deliver CBT to the patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT and computerized cognitive training (CCT) (Experimental): Participants will play CCT games at home 5 times per week for two weeks before beginning CBT and for two weeks after the first CBT session. Then participants will have CCT games immediately prior to CBT for nine more weeks (one time a week).
  Interventions: Behavioral: Cognitive behavioral therapy (CBT); Behavioral: computerized cognitive training (CCT)
- Cognitive behavioral therapy (Active Comparator): Participants will receive CBT sessions once a week for 12 weeks.
  Interventions: Behavioral: Cognitive behavioral therapy (CBT)

INTERVENTIONS:
Behavioral: Cognitive behavioral therapy (CBT) — The CBT intervention will consist of 12 weekly 60 minute sessions of the manualized therapy, adapted from the Coping Cat program, for the treatment of pediatric anxiety disorders.
Behavioral: computerized cognitive training (CCT) — CCT intervention will consist of approximately 30 minutes of CCT games prior to each CBT session, to engage cognitive control capacity prior to receipt of CBT. The CCT games will be designed to target focused attention, response inhibition, working memory and multiple simultaneous attention to constitute a general executive function training, and activate neural systems associated with executive function/cognitive control. Difficulty of the games will be titrated individually and by session to avoid boredom and progressively activate the functional systems underlying cognitive control.
  Arms: CBT and computerized cognitive training (CCT)

SUMMARY:
This study will assign participants with anxiety to cognitive behavioral therapy (CBT) with computerized cognitive training (CCT). In addition, the study will have a control group and enroll age- and gender-matched anxious children assigned to CBT.

The hypothesis of this trial is that CCT with CBT will further increase task control network (TCN) activation and connectivity.

Both groups will have one CBT therapy session each week for 12 weeks. However, for participants in the CCT arm plus CBT they will also receive up to 4 weeks of at home CCT to complete during the two weeks prior to the first CBT session and during the two weeks after the first CBT session. CCT is to be done at home for approximately 30 minutes per day, 5 days per week. Additionally, participants in the CCT arm plus CBT will receive CCT for 30 minutes just prior to CBT sessions 4-12.

Each group will also have pre and post therapy functional magnetic resonance imaging (fMRI) and be asked to complete anxiety severity interviews and questionnaires throughout the study as well as after the treatment.

Update as of 4/7/2020: Enrollment and in-person-only interactions/interventions are temporarily paused due to COVID-19 and are expected to resume in the future. This is not a suspension of IRB approval.

Update as of 7/20/2020: Enrollment and in-person-only interactions/interventions are resumed.

ELIGIBILITY:
Inclusion Criteria:

* Parent or guardian willing to give informed consent, and children willing to give informed assent to participate in the study
* Must be actively enrolled and maintain eligibility in Dimensional Brain Behavior Predictors of CBT Outcomes in Pediatric Anxiety (HUM00118950; P.I. Fitzgerald) to participate in the study.

Exclusion Criteria:

* Color blindness

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-11-07 (Actual); Study Completion 2021-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yanni Liu, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CBT and Computerized Cognitive Training (CCT) | Cognitive Behavioral Therapy
Started | 6 | 15
Completed | 6 | 12
Not Completed | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Did not obtain second fMRI. | 0 | 1
Not completed — MRI failed/no second fMRI | 0 | 1

BASELINE CHARACTERISTICS:
Population: Because this is a per-protocol analysis, the data from the 3 participants who did not complete the trial were not included in the analysis.
Groups:
- Cognitive Behavioral Therapy (CBT) and Computerized Cognitive Training (CCT): Participants will play CCT games at home 5 times per week for two weeks before beginning CBT and for two weeks after the first CBT session. Then participants will have CCT games immediately prior to CBT for nine more weeks (one time a week).
  Cognitive behavioral therapy (CBT): The CBT intervention will consist of 12 weekly 60 minute sessions of the manualized therapy, adapted from the Coping Cat program, for the treatment of pediatric anxiety disorders.
  computerized cognitive training (CCT): CCT intervention will consist of approximately 30 minutes of CCT games prior to each CBT session, to engage cognitive control capacity prior to receipt of CBT. The CCT games will be designed to target focused attention, response inhibition, working memory and multiple simultaneous attention to constitute a general executive function training, and activate neural systems associated with executive function/cognitive control. Difficulty of the games will be titrated individually and by session to avoid boredom and progressively activate the functional systems underlying cognitive control.
- Cognitive Behavioral Therapy (CBT): Participants will receive CBT sessions once a week for 12 weeks.
  Cognitive behavioral therapy (CBT): The CBT intervention will consist of 12 weekly 60 minute sessions of the manualized therapy, adapted from the Coping Cat program, for the treatment of pediatric anxiety disorders.
- Participants Who Did Not Complete: Participants who were assigned to the Cognitive behavioral therapy arm, but who withdrew or did not complete the trial. Data from the participants in this arm was not included in the outcome measure data.
- Total: Total of all reporting groups
Arm/Group | Cognitive Behavioral Therapy (CBT) and Computerized Cognitive Training (CCT) | Cognitive Behavioral Therapy (CBT) | Participants Who Did Not Complete | Total
Number analyzed (Participants) | 6 | 12 | 3 | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.3 (3.6) | 12.4 (2.7) | 10.2 (1.0) | 12.6 (3.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 9 | 2 | 16
  Male | 1 | 3 | 1 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 9 | 3 | 16
  Multiracial: black/white/native | 1 | 0 | 0 | 1
  Multiracial: Bosniak | 0 | 1 | 0 | 1
  Multiracial: Caucasian/Asian | 0 | 1 | 0 | 1
  Other: Pacific Islander | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 12 | 3 | 21
Brain Activation and Connectivity in the Task-control Network (TCN) [Mean (Standard Deviation); unit: Arbitrary Units] — Population: During the fMRI scan, 1 participant in the "Participants Who Did Not Complete" arm moved too much. As a result, the participant's data was not usable.
  Because only 2 participants' data in the "Participants Who Did Not Complete" arm could be analyzed, the number of participants was too few to calculate a TCN for this arm, as correlation analysis required 3 or more participants' data.
  Arbitrary Units
    leftIFG: number analyzed (Participants) | 6 | 12 | 2 | 20
    leftIFG | 0.66 (0.180) | 0.696 (0.421) | 0.169 (0.258) | 0.612 (0.369)
    rightIFG: number analyzed (Participants) | 6 | 12 | 2 | 20
    rightIFG | 0.739 (0.423) | 0.801 (.798) | 0.428 (1.209) | 0.720 (0.694)
    leftParietal: number analyzed (Participants) | 6 | 12 | 2 | 20
    leftParietal | -0.002 (0.586) | 0.066 (0.576) | 0.659 (0.064) | 0.058 (0.591)
    rightParietal: number analyzed (Participants) | 6 | 12 | 2 | 20
    rightParietal | 1.037 (0.356) | 0.679 (0.605) | 1.038 (1.296) | 0.791 (0.614)
    leftdACC: number analyzed (Participants) | 6 | 12 | 2 | 20
    leftdACC | 0.876 (0.310) | 0.681 (0.418) | 0.607 (0.664) | 0.705 (0.410)
    rightdACC: number analyzed (Participants) | 6 | 12 | 2 | 20
    rightdACC | 0.997 (0.489) | 1.026 (0.719) | 0.678 (0.720) | 0.971 (0.612)
    leftInsula: number analyzed (Participants) | 6 | 12 | 2 | 20
    leftInsula | 0.535 (0.099) | 0.438 (0.379) | 0.086 (0.345) | 0.416 (0.325)
    rightInsula: number analyzed (Participants) | 6 | 12 | 2 | 20
    rightInsula | 0.73 (0.289) | 0.573 (0.41) | 0.433 (1.141) | 0.571 (0.463)
    TCN: number analyzed (Participants) | 6 | 12 | 2 | 20
    TCN | 0.20 (0.51) | 0.50 (0.24) | NA (NA) — TCN was based on a correlation analysis, which would require 3 or more participants' data to calculate. | 0.50 (0.23)
Pediatric Anxiety Rating Score (PARS) [Mean (Standard Deviation); unit: Score on a Scale] — This is a 50 question interview-based tool used to assess for the presence and severity of anxiety symptoms in children and adolescents utilizing parental and youth input to guide clinician ratings. The total scores on this scale range from 0 to 30, with scores above 13 indicating clinically meaningful anxiety.
  Score on a Scale | 12.5 (3.3) | 19.2 (2.6) | 17.7 (3.1) | 17.4 (3.8)
Conflict Task Reaction Times [Mean (Standard Deviation); unit: milliseconds] — Population: During the fMRI scan, 1 participant in the "Participants Who Did Not Complete" arm moved too much. As a result, the participant's data was not usable.
  milliseconds
    number analyzed (Participants) | 6 | 12 | 2 | 20
    (all) | 800.8 (365.5) | 885.9 (256.7) | 1164.2 (421.2) | 888.2 (305)
Conflict Task Accuracy [Mean (Standard Deviation); unit: Percentage of correct responses] — Population: During the fMRI scan, 1 participant in the "Participants Who Did Not Complete" arm moved too much. As a result, the participant's data was not usable.
  Percentage of correct responses
    number analyzed (Participants) | 6 | 12 | 2 | 20
    (all) | 91 (3) | 86 (7) | 92.2 (1) | 88.3 (6)
NIH Toolbox Composite Score [Mean (Standard Deviation); unit: T-score] — An app-based cognitive assessment of executive function, attention, memory, and language. The NIH toolbox standard score has a mean of 100 and standard deviation (SD) of 15. The higher the score, the better the performance. Population: Data for 2 participants in the Participants Who Did Not Complete arm was collected but was rendered unusable because of technical difficulties.
  T-score
    number analyzed (Participants) | 6 | 12 | 1 | 19
    (all) | 111.2 (4.8) | 101.9 (11.4) | 106 | 105.0 (10.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Brain Activation and Connectivity in the Task-control Network (TCN)
Description: Pre- to post-CBT changes in brain activation and function connectivity in the task-control network including fronto-parietal and cingulo-opercular regions mediating cognitive control. Functional activation and connectivity of these brain regions are assessed using a conflict interference computer task performed during MRI scanning.
Time Frame: Baseline, 12 weeks (after therapy)
Population: One participant's fMRI data in the Cognitive Behavioral Therapy arm was not usable.
Measure: Mean (Standard Deviation); unit: Arbitrary Units
Arm/Group | CBT and Computerized Cognitive Training (CCT) | Cognitive Behavioral Therapy
Number analyzed (Participants) | 6 | 11
Arbitrary Units
  leftIFG (Change in Brain activity [post minus pre]) | 0.020 (0.151) | -0.206 (0.561)
  rightIFG (Change in Brain activity [post minus pre]) | 0.305 (0.742) | -0.004 (0.653)
  leftParietal (Change in Brain activity [post minus pre]) | 0.082 (0.095) | -0.096 (0.559)
  rightParietal (Change in Brain activity [post minus pre]) | -0.356 (0.375) | -0.032 (0.66)
  leftdACC (Change in Brain activity [post minus pre]) | -0.246 (0.26) | 0.164 (0.405)
  rightdACC (Change in Brain activity [post minus pre]) | -0.203 (0.909) | -0.270 (1.069)
  leftInsula (Change in Brain activity [post minus pre]) | -0.221 (0.399) | 0.081 (0.388)
  rightInsula (Change in Brain activity [post minus pre]) | -0.166 (0.541) | 0.067 (0.702)
  TCN (Change in Connectivity [post minus pre]) | 0.20 (0.47) | 0.53 (0.26)
Statistical Analysis 1: Comparison: CBT and Computerized Cognitive Training (CCT) vs Cognitive Behavioral Therapy; leftIFG (Change in Brain activity [post minus pre]); Test type: Superiority; Mean Difference (Final Values) = -0.226
Statistical Analysis 2: Comparison: CBT and Computerized Cognitive Training (CCT) vs Cognitive Behavioral Therapy; rightIFG (Change in Brain activity [post minus pre]); Test type: Superiority; Median Difference (Final Values) = -0.309
Statistical Analysis 3: Comparison: CBT and Computerized Cognitive Training (CCT) vs Cognitive Behavioral Therapy; leftParietal (Change in Brain activity [post minus pre]); Test type: Superiority; Mean Difference (Final Values) = -0.179
Statistical Analysis 4: Comparison: CBT and Computerized Cognitive Training (CCT) vs Cognitive Behavioral Therapy; rightParietal (Change in Brain activity [post minus pre]); Test type: Superiority; Mean Difference (Final Values) = 0.324
Statistical Analysis 5: Comparison: CBT and Computerized Cognitive Training (CCT) vs Cognitive Behavioral Therapy; leftdACC (Change in Brain activity [post minus pre]); Test type: Superiority; Mean Difference (Final Values) = 0.410
Statistical Analysis 6: Comparison: CBT and Computerized Cognitive Training (CCT) vs Cognitive Behavioral Therapy; rightdACC (Change in Brain activity [post minus pre]); Test type: Superiority; Mean Difference (Final Values) = -0.067
Statistical Analysis 7: Comparison: CBT and Computerized Cognitive Training (CCT) vs Cognitive Behavioral Therapy; leftInsula (Change in Brain activity [post minus pre]); Test type: Superiority; Mean Difference (Final Values) = 0.302
Statistical Analysis 8: Comparison: CBT and Computerized Cognitive Training (CCT) vs Cognitive Behavioral Therapy; rightInsula (Change in Brain activity [post minus pre]); Test type: Superiority — rightInsula (Change in Brain activity [post minus pre]); Mean Difference (Final Values) = 0.234
Statistical Analysis 9: Comparison: CBT and Computerized Cognitive Training (CCT) vs Cognitive Behavioral Therapy; TCN (Change in Connectivity [post minus pre]); Test type: Superiority; Mean Difference (Final Values) = -0.040

2. Secondary Outcome: Change in Pediatric Anxiety Rating Score (PARS)
Description: This is a 50-question interview-based tool used to assess for the presence and severity of anxiety symptoms in children and adolescents utilizing parental and youth input to guide clinician ratings. The total scores on this scale range from 0 to 30, with scores above 13 indicating clinically meaningful anxiety. The numbers presented represent the value at 12 weeks minus the value at baseline
Time Frame: Baseline, 12 weeks (after therapy)
Population: Data for 2 participants in the "CBT and computerized cognitive training (CCT)" arm are missing.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | CBT and Computerized Cognitive Training (CCT) | Cognitive Behavioral Therapy
Number analyzed (Participants) | 4 | 12
score on a scale | -5 (6.8) | -7.1 (4.4)
Statistical Analysis 1: Comparison: CBT and Computerized Cognitive Training (CCT) vs Cognitive Behavioral Therapy; Test type: Superiority; p = 0.241, t-test, 1 sided

3. Secondary Outcome: Change in Behavioral Performance on the Conflict Interference Task- Conflict Task Reaction Times
Description: Pre- to post-CBT changes in the behavioral performance in a conflict interference task. The time for the task at 12 weeks minus at baseline yields a number whose absolute value of change is shown below. Thus, when assessing the change, the higher number corresponds to more improvement in reaction time.
Time Frame: Baseline, 12 weeks (after therapy)
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | CBT and Computerized Cognitive Training (CCT) | Cognitive Behavioral Therapy
Number analyzed (Participants) | 6 | 12
milliseconds | 27.4 (55.3) | 70.7 (135)
Statistical Analysis 1: Comparison: CBT and Computerized Cognitive Training (CCT) vs Cognitive Behavioral Therapy; Test type: Superiority; p = 0.233, t-test, 1 sided

4. Secondary Outcome: Change in Behavioral Performance on the Conflict Interference Task- Conflict Task Accuracy
Description: Pre- to post-CBT changes in the behavioral performance in a conflict interference task. Conflict interference task refers to a task assigned to a participant to complete that also includes some form of distraction or condition that interferes with completion of the task. For this, the lower number indicates more improvement in accuracy in competing the task.
Time Frame: Baseline, 12 weeks (after therapy)
Measure: Mean (Standard Deviation); unit: percentage of correct responses
Arm/Group | CBT and Computerized Cognitive Training (CCT) | Cognitive Behavioral Therapy
Number analyzed (Participants) | 6 | 12
percentage of correct responses | -4.6 (3.6) | 9 (6.8)
Statistical Analysis 1: Comparison: CBT and Computerized Cognitive Training (CCT) vs Cognitive Behavioral Therapy; Test type: Superiority; p = 0.042, t-test, 1 sided

5. Secondary Outcome: Change in Tasks Testing Cognitive Control Capacity Included in the NIH Toolbox
Description: Pre- to post-CBT changes in the NIH toolbox composite score from the cognitive control module included in the toolbox. The NIH toolbox standard score has a mean of 100 and standard deviation (SD) of 15. The lower the change in the score between the pre- and the post-CBT changes indicates the higher degree of improvement.
Time Frame: Baseline, 12 weeks (after therapy)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | CBT and Computerized Cognitive Training (CCT) | Cognitive Behavioral Therapy
Number analyzed (Participants) | 6 | 12
T-score | -6.6 (10.7) | -8.4 (7.8)
Statistical Analysis 1: Comparison: CBT and Computerized Cognitive Training (CCT) vs Cognitive Behavioral Therapy; Test type: Superiority; p = 0.349, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | CBT and Computerized Cognitive Training (CCT) | Cognitive Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/15
Other Adverse Events (participants affected / at risk) | 0/6 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT04157296/Prot_SAP_001.pdf
  • Informed Consent Form (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/96/NCT04157296/ICF_000.pdf